CLINICAL TRIAL: NCT00822211
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study to Compare the Effect of 24 Weeks Treatment With Vildagliptin 50 mg Bid to Placebo as Add-On Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy
Brief Title: Efficacy of add-on Therapy With Vildagliptin in Chinese Patients With Type 2 Diabetes Inadequately Controlled With Prior Metformin Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23140
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; HbA1c reduction; vildagliptin; add-on to metformin; Chinese patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vildagliptin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Vildagliptin Dose 1 (Experimental)
  Interventions: Drug: Vildagliptin 50 mg bid
- Vildagliptin Dose 2 (Experimental)
  Interventions: Drug: Vildagliptin 50 mg qd
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin 50 mg bid
  Arms: Vildagliptin Dose 1
Drug: Vildagliptin 50 mg qd
  Arms: Vildagliptin Dose 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of vildagliptin 50 mg bid compared to placebo as an add-on therapy to metformin in Chinese patients with T2DM inadequately controlled by metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM who have received metformin for at least 8 weeks and have been on a stable dose of at least 1500 mg daily for a minimum of 4 weeks prior to visit 1
* Agreement to maintain the same dose of metformin from randomization to the end of the study
* Age in the range of 18-78 years inclusive
* Body mass index (BMI) in the range of 20-40 kg/m2 inclusive at Visit 1
* HbA1c in the range of > 7.0 to ≤10% at Visit 1
* Agreement to maintain prior diet and exercise habits during the full course of the study
* Ability to comply with all study requirements

Exclusion Criteria:

* Fasting Plasma Glucose (FPG) > 270 mg/dl (15 mmol/L) at Visit 1
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c after 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Percent of patients with HbA1c < 7% after 24 weeks | 24 weeks
Adverse event profile after 24 weeks of treatment | 24 weeks
Change from baseline in fasting plasma glucose at 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- China (17):
  - China-Japan Friendship Hospital, Beijing
  - General Hospital of Beijing Military Region of PLA, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - The General Hospital of the PLA, Beijing
  - The General Hospital of the Second Artilleryman of PLA, Beijing
  - The Affiliated Union Hospital of Fujian Medical University, Fuzhou
  - The Fuzhou General Hospital of the PLA Nanjing Military Area, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Second Affiliated Hospital of Nanchang University, Nanchang
  - The Jiangxi Provincial People's Hospital, Nanchang
  - Te Affiliated Drum Tower of Nanjing University Medical School, Nanjing
  - Tongji Hospital of Tongji University, Nanjing
  - Shanghai Changzheng Hospital, Shanghai
  - The Second Affiliated Hospital of China Medical University, Shenyang
  - The Second Affiliated Hospital of Tianjin Medical University, Tianjin
  - First Affiliated Hospital of 4th Military Medical University, Xi'an

REFERENCES:
- [Result] Pan C, Xing X, Han P, Zheng S, Ma J, Liu J, Lv X, Lu J, Bader G; Institution Investigators. Efficacy and tolerability of vildagliptin as add-on therapy to metformin in Chinese patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2012 Aug;14(8):737-44. doi: 10.1111/j.1463-1326.2012.01593.x. Epub 2012 Apr 1. PMID 22369287